CLINICAL TRIAL: NCT05397314
Title: DNA Fragmentation - Effect on Pregnancy Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jens Fedder, Professor, Odense University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: S-20140212
Record Dates: First submitted 2019-10-15; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Punalpin (Experimental)
  Interventions: Dietary Supplement: Punalpin
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Punalpin
  Arms: Punalpin
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Punalpin, an antioxidant, has a positive impact on DNA fragmentation in spermatozoa in male fertility patients with increased amount of DNA fragmentation in their spermatozoa. Secondary purpose is to investigate whether there is any positive effect on the subsequent pregnancy rates from the fertility treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male fertility patients with increased amount of DNA fragmentation in their spermatozoa

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-01-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Sperm DNA fragmentation | 4 months
  Reduction in DNA fragmentation